CLINICAL TRIAL: NCT05291013
Title: Adipose Tissue Dysfunction in Type 2 Diabetes and Its Reversibility by Bariatric Surgery
Acronym: ADIDYS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Kristoffer Jensen Kolnes, MD, PhD-student, Odense University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20190162
Record Dates: First submitted 2022-03-14; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Adipose Tissue Dysfunction Type 2 Diabetes Mellitus Bariatric Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gastric bypass with T2DM (Experimental)
  Interventions: Procedure: Gastric byspass
- Gastric bypass without T2DM (Experimental)
  Interventions: Procedure: Gastric byspass
- Control group (No Intervention)

INTERVENTIONS:
Procedure: Gastric byspass — Test will be before and 9-12 month after gastric bypass
  Arms: Gastric bypass with T2DM; Gastric bypass without T2DM

SUMMARY:
ABSTRACT Background: Insulin resistance (IR) plays a major role in the pathogenesis of type 2 diabetes (T2D). Adipose tissue (AT) dysfunction leading to systemic low-grade inflammation and ectopic lipid deposition plays an important role in obesity-induced IR, but its role in T2D pathogenesis and to what extent insulin-sensitizing interventions can reverse AT dysfunction remain to be clarified.

Hypothesis/aims: To test the hypotheses 1) that T2D is associated with exaggerated AT dysfunction compared with obesity alone, 2) that increased insulin sensitivity and remission of T2D after bariatric surgery is in part explained by improved AT function Research plan: Novel markers of exaggerated AT dysfunction will be identified and studied together with known markers of AT dysfunction in patients with T2D compared with non-diabetic obese and lean individuals. Then the effects of bariatric surgery on all these markers of AT dysfunction in obesity and T2D will be studied. Adipose tissue and skeletal muscle biopsies and blood samples will be used for 1) next generation RNA sequencing, 2) targeted analysis of mRNA and protein content/activities, 3) metabolomics, 4) morphological analysis and 5) analysis of adipokines/myokines. Abnormalities in T2D and changes in response to bariatric surgery will be related to substrate metabolism, insulin sensitivity and secretion and insulin signalling in muscle.

Perspectives: This project provides novel insight into the role of AT dysfunction in T2D pathogenesis in humans and the potential of bariatric surgery to reverse AT dysfunction and improve insulin sensitivity. We ultimately expect that this will help us to identify novel pharmaceutical targets for the treatment of IR.

ELIGIBILITY:
Inclusion Criteria:

* GAD65 antibody negative patients with T2D
* Treated with either diet alone or diet in combination with metformin, DPP-4 inhibitors, sulphonylureas, GLP1-analogs or insulin (maximum 40 IE long - or intermediate acting insulin).
* HbA1c < 70 mmol/l for diabetics and <48 mmol/l for obese.
* Do not have any known diabetic complication (macroalbuminuria, proliferative retinopathy, neuropathy or cardiovascular disease).
* The use of up to two antihypertensive drugs and one cholesterol lowering drug is allowed in patients with T2D and obese individuals.
* Both patients with T2D and obese individuals should be eligible for bariatric surgery, and should be able and willing to discontinue all drugs for 1 week prior to the clamp studies
* Except for the conditions mentioned above, the patients with T2D and the obese individuals should be healthy.
* Lean controls should be healthy, lean and drug naive.
* Obese and lean controls should have no first degree family history of diabetes.
* All participants should be 30-65 years old.
* All participants should be able to provide informed written consent.

Exclusion Criteria:

* Any unknown disease or need for medication that occurs after inclusion.
* Abnormal ECG, screening blood tests and/or severe hypertension (>160/100 mmHg).
* Impaired glucose tolerance (IGT) or impaired fasting glucose in lean, healthy participants (2-hour plasma glucose > 7.8 mmol/l or fasting plasma glucose > 5.6 mmol/l).
* Known pregnancy or positive beta-HCG in blood during screening.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Markers in adipose tissue dysfunction | 3 year
  Changes in morphology of adipocytes, mRNA expression and protein abundance in adipocytes
Muscular insulin sensitivity | 3 year
  Changes in muscle mRNA expression and protein abundance

SECONDARY OUTCOMES:
Rate of disposal | 3 year
  Changes in rate of disposal
Body composition | 3 year
  Changes in body composition
Metabolomics | 3 year
  Changes in metabolomics

CONTACTS AND LOCATIONS:
Locations (1):
- Kristoffer Jensen Kolnes, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided